CLINICAL TRIAL: NCT02539030
Title: Random Clinical Trial for Comparison of Efficacy and Safety of Simple Microfracture and Modified Microfracture Using Collagen in the Patients With Knee Cartilage Defects
Brief Title: Comparison of Efficacy and Safety of Microfracture and Modified Microfracture
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03CAR
Record Dates: First submitted 2015-08-28; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Defect of Articular Cartilage; Osteoarthritis; Traumatic Arthritis
Keywords: Cartilage defect of knee; microfracture; modified microfracture; collagen
MeSH Terms: conditions — Osteoarthritis; Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- microfracture (Active Comparator): simple microfracture for cartilage defect of knee
  Interventions: Procedure: Microfracture
- modified microfracture using collagen (Experimental): modified microfracture using collagen (CartiFill) for cartilage defect of knee
  Interventions: Procedure: Microfracture; Device: CartiFill

INTERVENTIONS:
Procedure: Microfracture — simple microfracture
Device: CartiFill — add collagen when doing microfracture
  Arms: modified microfracture using collagen

SUMMARY:
This study was designed to evaluate the efficacy and safety of a modified microfracture using collagen, and to compare them with those of a simple microfracture to prove the non-inferiority of the modified microfracture using collagen in patients with cartilage defects in their knees.

DETAILED DESCRIPTION:
This study was an open-trial study. One hundred subjects participated in it. The study was explained to the subjects and they voluntarily agreed to participate in it. Their eligibility to participate in the study was checked, and they were randomized either into the simple microfracture group or the modified microfracture group using collagen based on a centrally controlled randomization table. They were asked to follow the guidelines of the investigators during the study and to visit the hospital six times*, including for screening. At each visit, the subjects underwent an examination with doctors, a blood test, an X-ray procedure, an MRI, an observation with the naked eyes, and arthroscopy to evaluate the safety and efficacy of the procedure. (*If the screening date overlaps with the procedure date, the number of his or her visits would be five.)

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with cartilage defects in their knee (Including Knee OA and Knee TA) 2. Knee osteoarthritis patients whose Kellgren-Lawrence Grading Scale score is lower than 3 (patients who received simultaneous or previous correction will be excluded).

3. Patients with misalignment of their tibia and femur, unstable ligament in their knee, or bony defects in the lesions of their knee, and/or who had been treated for alignment 4. Patients who were 15 years old or older 5. Patients or their representative (for adults), or patients and their parent/guardian (for minors), who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

* 1. If patients or their families suffer from or have ever suffered from an autoimmune disease.

  2. Patients who have ever suffered an anaphylactic reaction. 3. Patients who have ever suffered hypersensitivity to an implant. 4. Patients with a history of allergy to porcine or bovine protein. 5. Subjects with inflammatory arthritis, such as rheumatoid and gouty arthritis.

  6. Subjects with autoimmune disease related arthritis. 7. Subjects who are pregnant and/or breast-feeding and/or plan a pregnancy. 8. Subjects with tumors. 9. Subjects who have undergone radiotherapy or chemotherapy within the last 2 years (Exception: if the possibility of collagen treatment is confirmed with doctor's clinical decision).

  10. Subjects who are diabetic. (Exception: if the possibility of CartiFill™ treatment is confirmed with doctor's clinical decision, and/or patient's blood glucose level remains within the normal range and/or no other complications by diabetes mellitus.) 11. Subjects with infections, currently on treatment with antibiotics or antimicrobials (Exception: if the possibility of collagen treatment is confirmed with doctor's clinical decision).

  12. Subjects under adrenocorticoid therapy (Exception: if the possibility of collagen treatment is confirmed with doctor's clinical decision).

  13. Subjects with psychiatric disorders who are considered inappropriate to participate in this trial by the Principal Investigator.

  14. Patients who have ever suffered contraindications of the used Fibrin sealant. (The major contraindications are as follows: patients with hypersensitivity to aprotinin and those treatments for severe brisk arterial or venous bleeding.)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
100mmVAS(Visual Analogue Scale) | 12 month after surgery
  It will be evaluated by the VAS score 12 months after surgery of the affected knee of the investigational group and the control group.

SECONDARY OUTCOMES:
change of 100 mmVAS (Visual Analogue Scale) | screening, 3, 6, 12 and 24 months after surgery
  The difference between the VAS scores of the affected knee at the screening and 12 months after surgery in the investigational group will be compared to that in the control group. The differences in the VAS scores obtained at the follow-ups (3, 6, and 24 months after surgery) will be compared.
change of Knee injury and osteoarthritis outcome (KOOS) | screening, 6, 12 and 24 months after surgery
  The difference between the KOOS scores of the affected knee at the screening and 12 months after surgery in the investigational group will be compared to that in the control group. The differences in the KOOS scores obtained at the follow-ups (6 and 24 months after surgery) will be compared.
change of International Knee Documentation Committee (IKDC) | screening, 6, 12 and 24 months after surgery
  The difference between the IKDC scores of the affected knee at the screening and 12 months after the surgery in the investigation group will be compared to that in the control group. The differences in the IKDC scores obtained at the follow-ups (6 and 24 months after surgery) will be compared.
the results of MRI and MRI of articular cartilage examination (T2, T2 star, deGEMRIC, UTE, etc.), mMOCART | 12 months after surgery
  The results obtained 12 months after the surgery on the affected knee in the investigational and control groups will be described. mMOCART will be obtained, and the difference will be assessed.
  * Depending on the MRI equipment, if in-house imaging is not possible, it may be done at the other hospitals conducting the research.

CONTACTS AND LOCATIONS:
Overall Officials: Nam Yong Choi, MD, Principal Investigator — Catholic University of Korea Saint Paul's Hospital; Yong In, MD, Principal Investigator — The Catholic University of Korea; Chan Woong Moon, MD, Principal Investigator — The Catholic University of Korea Bucheon St.Mary's Hospital; Hae Seock Ko, MD, Principal Investigator — The Catholic University of Korea Vincent's Hospital; Cheol Hong Jeon, MD, Principal Investigator — Wonkwang University Hospital; Seung Back Kang, MD, Principal Investigator — SMG-SNU Boramae Medical Center; Ja Young Choi, MD, Principal Investigator — Seoul National University Hospital; Myung Koo Kim, MD, Principal Investigator — Inha University Hospital; Jae Kyun Jun, MD, Principal Investigator — Daejeon Sun hospital; Jae Doo Yoo, MD, Principal Investigator — Ewha Womans University Mokdong Hospital; Jung Koo Ha, MD, Principal Investigator — Inje University; Jun Ho Wang, MD, Principal Investigator — Samsung Medical Center
Locations (12):
- South Korea (12):
  - Daejeon Sun hospital, Daejeon, Daejeon
  - The Catholic University of Korea Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea Vincent's Hospital, Suwon, Gyeonggi-do
  - Inha University Hospital, Incheon, Incheon
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul
  - Inje University Seoul Paik Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, Seoul
  - Seoul National University Hospital, Seoul, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Seoul
  - The Catholic University of Korea St. Paul's Hospital, Seoul, Seoul

REFERENCES:
- [Derived] Kim MS, Chun CH, Wang JH, Kang SB, Chang MJ, In Y. Microfracture Versus a Porcine-Derived Collagen-Augmented Chondrogenesis Technique for Treating Knee Cartilage Defects: Results at Midterm Follow-up. Orthop J Sports Med. 2024 Nov 7;12(11):23259671241292093. doi: 10.1177/23259671241292093. eCollection 2024 Nov. PMID 39525351